CLINICAL TRIAL: NCT03350854
Title: An Intervention to Improve Decision Role Concordance Amongst Newly Diagnosed Breast Cancer Patients
Brief Title: Improving Decision Role Concordance in Newly Diagnosed Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Cindy Matsen, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB_00081898
Record Dates: First submitted 2017-10-13; First posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer
Keywords: early stage breast cancer;; treatment decision making; newly diagnosed breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The non-intervention control group (No Intervention): In the non-intervention control group, providers are blind to the patient's preferred decision making role.
- The intervention group (Experimental): The provider will be informed of the patient preference in treatment decision making (preferred role) and have a discussion about this with the patient in the intervention group.
  Interventions: Behavioral: Patient Preference in Treatment Decision Making

INTERVENTIONS:
Behavioral: Patient Preference in Treatment Decision Making — The roles are divided into two active roles, a collaborative (or shared) role, and two passive roles in the Patient Preference scale questionnaire. Once the questionnaire is administered, the patient will then proceed to original surgical appointment. The provider is informed of the patient's preferred role and has a discussion with them patient about this in the intervention group, but not in the control group.
  Arms: The intervention group

SUMMARY:
The goal of this project is to test the effects of the Patient Preference Scale as the basis for a clinical intervention for role negotiation in breast cancer surgery decisions and the Patient Perception Scale to measure role concordance. The investigators hypothesize that better role concordance will be achieved with a simple provider-based intervention. In the first half of the study, providers will be blind to the patient's preferred role. In the second half, providers will be made aware of the preferred role prior to the encounter and will have a brief conversation with the patient about their desired role in the decision making process.

DETAILED DESCRIPTION:
The goal of this project is to test the effects of the Patient Preference Scale as the basis for a clinical intervention for role negotiation in breast cancer surgery decisions and the Patient Perception Scale to measure role concordance. The investigators hypothesize that better role concordance will be achieved with a simple provider-based intervention. In addition, role concordance will be associated with improved short-term and longer-term improvements in outcomes of the following parameters: a) satisfaction with decision process b) breast specific QOL, and c) decision regret.

The investigators propose a mixed methods, interventional study with concurrent controls performed in a breast cancer surgery clinic at a comprehensive cancer center. The Patient Preference Scale will be used to identify the preferred involvement in decision making of newly diagnosed breast cancer patients prior to their first clinic visit. The Patient Perception Scale will be used after the encounter in order to evaluate role concordance. The Provider Perception Scale will also be used to assess the perception of the achieved role by the provider. In the first half of the study, providers will be blind to the patient's preferred role. In the second half, providers will be made aware of the preferred role prior to the encounter and will have a brief conversation with the patient about their desired role in the decision making process. Clinical encounters will be audiotaped, transcribed, and scored for patient involvement. The investigators propose the following aims and hypotheses:

Investigate the impact of a brief provider-led intervention about the patients' preferred role in treatment decision making on role concordance. The investigators hypothesize that:

1. Role concordance will be improved when the preferred role is discussed with the patient at the beginning of the encounter.

2. The provider's perception of the role achieved will be more concordant with the patient's perception when the preferred role is discussed. 3. Investigate the impact of role concordance in the treatment decision making process on short term and long term quality of life and decision outcomes. The investigators hypothesize that: Patients who achieve role concordance will be more satisfied with the decision process.

1. Patients who achieve role concordance will have better QOL and less decision regret at early (2 to 6 weeks) and later (6 months) time points after the clinic visit.
2. Patients who achieve concordance will be more likely to complete or plan to complete recommended treatments.
3. Patients who achieve concordance will be more likely to complete or plan to complete recommended treatments

ELIGIBILITY:
Inclusion Criteria:

* All patients who present to Huntsman Cancer Hospital/University of Utah for a newly diagnosed breast cancer surgical consultation.

Exclusion Criteria:

* Men with breast cancer.
* Patients who have previously seen another medical provider to discuss treatment for newly diagnosed breast cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is based on gender (female breast cancer patients)
Enrollment: 100 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-08-09 (Actual)

PRIMARY OUTCOMES:
Decision role concordance before and after a surgical consultation | The estimated period is 3 hours (before and immediately after a surgical consultation)
  The primary outcome measures the changes from patient's preferred role in baseline (before a surgical consultation) to the perception of whether the patient achieved the preferred role (immediately after a surgical consultation) in the surgical consultation.
Decision role concordance of provider and patient | This is an one-time measurement (Immediately after a surgical consultation)
  It measures the difference in the patient's perception of the achieved role and provider's perception of the patient's preferred role.

SECONDARY OUTCOMES:
Patient's satisfaction with the decision making process | immediately after a surgical consultation
  Satisfaction with the decision making process will be measured directly after the clinic encounter using a modified version of the Holmes-Rovner Satisfaction with Decision scale. The scale uses a Likert-type ranking of 6 items related to decision making, with 1 being strongly disagree and 5 being strongly agree.
Comparing Reliability and Validity of the Functional Assessment of Cancer Therapy-Breast (FACT-B) assessment of short-term quality of life between the groups | This scale will be used prior to the first consultation to establish a baseline for each patient and will subsequently be used at 2 weeks and 6 months after initial clinic visit.
  Quality of life will be assessed using the (FACT-B) questionnaire. FACT-B measures 27 items in five different areas: physical well-being, social/family well-being, emotional well-being, functional well-being, and additional concerns specific to this patient population. FACT-B is measured on the scale from 0 to 4, with a total minimum score of 0 and maximum score of 144.
The Decision Regret outcome | The scale will be administered at 2 weeks and 6 months after initial clinic visit.
  The decision regret outcome will be measured using the Decision Regret Scale. The Decision Regret Scale is is a 5 item scale with items ranked on a 5-point Likert-type scale and added together with higher score indicating more regret.
Observing Patient Involvement in Decision Making (OPTION) assessment of patient involvement | 4 months after initial clinic visit
  The outcome of patient involvement at the clinic encounter will be measured using the OPTION scale. This scale measures 12 item from 0 to 4, with 0 being "this behavior is not observed" to 4 "This behavior is exhibited to a very high standard"
completion or intention to complete therapies | 6 months after initial clinic visit
  Group differences in completion or intention to complete recommended therapies will be assessed at 6 months after the clinic visit through chart review of all participants' charts.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Matsen, MD, Principal Investigator — University of Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sepucha K, Ozanne EM. How to define and measure concordance between patients' preferences and medical treatments: A systematic review of approaches and recommendations for standardization. Patient Educ Couns. 2010 Jan;78(1):12-23. doi: 10.1016/j.pec.2009.05.011. Epub 2009 Jun 30. PMID 19570647
- [Background] Sepucha KR, Barry MJ. Making patient-centered cancer care a reality. Cancer. 2009 Dec 15;115(24):5610-1. doi: 10.1002/cncr.24824. No abstract available. PMID 19957353
- [Background] Dwamena F, Holmes-Rovner M, Gaulden CM, Jorgenson S, Sadigh G, Sikorskii A, Lewin S, Smith RC, Coffey J, Olomu A. Interventions for providers to promote a patient-centred approach in clinical consultations. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD003267. doi: 10.1002/14651858.CD003267.pub2. PMID 23235595
- [Background] Stiggelbout AM, Pieterse AH, De Haes JC. Shared decision making: Concepts, evidence, and practice. Patient Educ Couns. 2015 Oct;98(10):1172-9. doi: 10.1016/j.pec.2015.06.022. Epub 2015 Jul 15. PMID 26215573
- [Background] Livaudais JC, Franco R, Fei K, Bickell NA. Breast cancer treatment decision-making: are we asking too much of patients? J Gen Intern Med. 2013 May;28(5):630-6. doi: 10.1007/s11606-012-2274-3. Epub 2012 Nov 15. PMID 23229908
- [Background] Katz SJ, Lantz PM, Janz NK, Fagerlin A, Schwartz K, Liu L, Deapen D, Salem B, Lakhani I, Morrow M. Patient involvement in surgery treatment decisions for breast cancer. J Clin Oncol. 2005 Aug 20;23(24):5526-33. doi: 10.1200/JCO.2005.06.217. PMID 16110013
- [Background] Chewning B, Bylund CL, Shah B, Arora NK, Gueguen JA, Makoul G. Patient preferences for shared decisions: a systematic review. Patient Educ Couns. 2012 Jan;86(1):9-18. doi: 10.1016/j.pec.2011.02.004. Epub 2011 Apr 6. PMID 21474265
- [Background] Singh JA, Sloan JA, Atherton PJ, Smith T, Hack TF, Huschka MM, Rummans TA, Clark MM, Diekmann B, Degner LF. Preferred roles in treatment decision making among patients with cancer: a pooled analysis of studies using the Control Preferences Scale. Am J Manag Care. 2010 Sep;16(9):688-96. PMID 20873956
- [Background] Frongillo M, Feibelmann S, Belkora J, Lee C, Sepucha K. Is there shared decision making when the provider makes a recommendation? Patient Educ Couns. 2013 Jan;90(1):69-73. doi: 10.1016/j.pec.2012.08.016. Epub 2012 Sep 20. PMID 22999786
- [Background] Degner LF, Sloan JA, Venkatesh P. The Control Preferences Scale. Can J Nurs Res. 1997 Fall;29(3):21-43. PMID 9505581
- [Background] Degner LF, Kristjanson LJ, Bowman D, Sloan JA, Carriere KC, O'Neil J, Bilodeau B, Watson P, Mueller B. Information needs and decisional preferences in women with breast cancer. JAMA. 1997 May 14;277(18):1485-92. PMID 9145723
- [Background] Janz NK, Wren PA, Copeland LA, Lowery JC, Goldfarb SL, Wilkins EG. Patient-physician concordance: preferences, perceptions, and factors influencing the breast cancer surgical decision. J Clin Oncol. 2004 Aug 1;22(15):3091-8. doi: 10.1200/JCO.2004.09.069. PMID 15284259
- [Background] Tariman JD, Berry DL, Cochrane B, Doorenbos A, Schepp K. Preferred and actual participation roles during health care decision making in persons with cancer: a systematic review. Ann Oncol. 2010 Jun;21(6):1145-1151. doi: 10.1093/annonc/mdp534. Epub 2009 Nov 25. PMID 19940010
- [Background] Johnson JD, Roberts CS, Cox CE, Reintgen DS, Levine JS, Parsons M. Breast cancer patients' personality style, age, and treatment decision making. J Surg Oncol. 1996 Nov;63(3):183-6. doi: 10.1002/(SICI)1096-9098(199611)63:33.0.CO;2-9. PMID 8944063
- [Background] Almyroudi A, Degner LF, Paika V, Pavlidis N, Hyphantis T. Decision-making preferences and information needs among Greek breast cancer patients. Psychooncology. 2011 Aug;20(8):871-9. doi: 10.1002/pon.1798. Epub 2010 Jul 11. PMID 20623805
- [Background] Budden LM, Pierce PF, Hayes BA, Buettner PG. Australian women's prediagnostic decision-making styles, relating to treatment choices for early breast cancer treatment. Res Theory Nurs Pract. 2003 Summer;17(2):117-36. doi: 10.1891/rtnp.17.2.117.53178. PMID 12880217
- [Background] Vogel BA, Bengel J, Helmes AW. Information and decision making: patients' needs and experiences in the course of breast cancer treatment. Patient Educ Couns. 2008 Apr;71(1):79-85. doi: 10.1016/j.pec.2007.11.023. Epub 2008 Jan 8. PMID 18191933
- [Background] Vogel BA, Helmes AW, Hasenburg A. Concordance between patients' desired and actual decision-making roles in breast cancer care. Psychooncology. 2008 Feb;17(2):182-9. doi: 10.1002/pon.1215. PMID 17534866
- [Background] Wallberg B, Michelson H, Nystedt M, Bolund C, Degner LF, Wilking N. Information needs and preferences for participation in treatment decisions among Swedish breast cancer patients. Acta Oncol. 2000;39(4):467-76. doi: 10.1080/028418600750013375. PMID 11041108
- [Background] Lantz PM, Janz NK, Fagerlin A, Schwartz K, Liu L, Lakhani I, Salem B, Katz SJ. Satisfaction with surgery outcomes and the decision process in a population-based sample of women with breast cancer. Health Serv Res. 2005 Jun;40(3):745-67. doi: 10.1111/j.1475-6773.2005.00383.x. PMID 15960689
- [Background] Hack TF, Pickles T, Ruether JD, Weir L, Bultz BD, Mackey J, Degner LF. Predictors of distress and quality of life in patients undergoing cancer therapy: impact of treatment type and decisional role. Psychooncology. 2010 Jun;19(6):606-16. doi: 10.1002/pon.1590. PMID 19557823
- [Background] Hack TF, Degner LF, Watson P, Sinha L. Do patients benefit from participating in medical decision making? Longitudinal follow-up of women with breast cancer. Psychooncology. 2006 Jan;15(1):9-19. doi: 10.1002/pon.907. PMID 15669023
- [Background] Hyphantis T, Almyroudi A, Paika V, Degner LF, Carvalho AF, Pavlidis N. Anxiety, depression and defense mechanisms associated with treatment decisional preferences and quality of life in non-metastatic breast cancer: a 1-year prospective study. Psychooncology. 2013 Nov;22(11):2470-7. doi: 10.1002/pon.3308. Epub 2013 May 27. PMID 23712915
- [Background] Hawley ST, Lillie SE, Morris A, Graff JJ, Hamilton A, Katz SJ. Surgeon-level variation in patients' appraisals of their breast cancer treatment experiences. Ann Surg Oncol. 2013 Jan;20(1):7-14. doi: 10.1245/s10434-012-2582-1. Epub 2012 Oct 6. PMID 23054105
- [Background] Gattellari M, Butow PN, Tattersall MH. Sharing decisions in cancer care. Soc Sci Med. 2001 Jun;52(12):1865-78. doi: 10.1016/s0277-9536(00)00303-8. PMID 11352412
- [Background] Keating NL, Guadagnoli E, Landrum MB, Borbas C, Weeks JC. Treatment decision making in early-stage breast cancer: should surgeons match patients' desired level of involvement? J Clin Oncol. 2002 Mar 15;20(6):1473-9. doi: 10.1200/JCO.2002.20.6.1473. PMID 11896094
- [Background] Hillyer GC, Hershman DL, Kushi LH, Lamerato L, Ambrosone CB, Bovbjerg DH, Mandelblatt JS, Rana S, Neugut AI. A survey of breast cancer physicians regarding patient involvement in breast cancer treatment decisions. Breast. 2013 Aug;22(4):548-54. doi: 10.1016/j.breast.2012.10.001. Epub 2012 Oct 27. PMID 23107518
- [Background] Nguyen F, Moumjid N, Charles C, Gafni A, Whelan T, Carrere MO. Treatment decision-making in the medical encounter: comparing the attitudes of French surgeons and their patients in breast cancer care. Patient Educ Couns. 2014 Feb;94(2):230-7. doi: 10.1016/j.pec.2013.07.011. Epub 2013 Dec 8. PMID 24325874
- [Background] de Haes H. Dilemmas in patient centeredness and shared decision making: a case for vulnerability. Patient Educ Couns. 2006 Sep;62(3):291-8. doi: 10.1016/j.pec.2006.06.012. Epub 2006 Jul 21. No abstract available. PMID 16859860
- [Background] Sivell S, Elwyn G, Edwards A, Manstead AS; BresDex group. Factors influencing the surgery intentions and choices of women with early breast cancer: the predictive utility of an extended theory of planned behaviour. BMC Med Inform Decis Mak. 2013 Aug 20;13:92. doi: 10.1186/1472-6947-13-92. PMID 23962230
- [Background] Fagerlin A, Lakhani I, Lantz PM, Janz NK, Morrow M, Schwartz K, Deapen D, Salem B, Liu L, Katz SJ. An informed decision? Breast cancer patients and their knowledge about treatment. Patient Educ Couns. 2006 Dec;64(1-3):303-12. doi: 10.1016/j.pec.2006.03.010. Epub 2006 Jul 24. PMID 16860523
- [Background] O'Leary KA, Estabrooks CA, Olson K, Cumming C. Information acquisition for women facing surgical treatment for breast cancer: influencing factors and selected outcomes. Patient Educ Couns. 2007 Dec;69(1-3):5-19. doi: 10.1016/j.pec.2007.08.002. Epub 2007 Sep 24. PMID 17889495
- [Background] Singer E, Couper MP, Fagerlin A, Fowler FJ, Levin CA, Ubel PA, Van Hoewyk J, Zikmund-Fisher BJ. The role of perceived benefits and costs in patients' medical decisions. Health Expect. 2014 Feb;17(1):4-14. doi: 10.1111/j.1369-7625.2011.00739.x. Epub 2011 Nov 10. PMID 22070416
- [Background] Sepucha K, Mulley AG Jr. A perspective on the patient's role in treatment decisions. Med Care Res Rev. 2009 Feb;66(1 Suppl):53S-74S. doi: 10.1177/1077558708325511. Epub 2008 Nov 10. PMID 19001081
- [Background] Street RL Jr, Elwyn G, Epstein RM. Patient preferences and healthcare outcomes: an ecological perspective. Expert Rev Pharmacoecon Outcomes Res. 2012 Apr;12(2):167-80. doi: 10.1586/erp.12.3. PMID 22458618
- [Derived] Gutnik L, Allen CM, Presson AP, Matsen CB. Breast Cancer Surgery Decision Role Perceptions and Choice of Surgery. Ann Surg Oncol. 2020 Oct;27(10):3623-3632. doi: 10.1245/s10434-020-08485-8. Epub 2020 Jun 3. PMID 32495282
- See also: AHRQ. National Healthcare Quality Report. 2005 [cited 2015 August 13] — http://archive.ahrq.gov/qual/nhqr05/nhqr05.htm

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-05-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT03350854/Prot_SAP_000.pdf
  • Informed Consent Form (2017-01-29): https://cdn.clinicaltrials.gov/large-docs/54/NCT03350854/ICF_001.pdf